CLINICAL TRIAL: NCT02347735
Title: Predictive Factors for Anastomotic Leakage After Colorectal Surgery: The REVEAL Study
Brief Title: Predictive Factors for Anastomotic Leakage After Colorectal Surgery
Acronym: REVEAL
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Zuyderland Medical Centre (Other); VieCuri Medical Centre (Other)
Responsible Party: Sponsor
Other Study IDs: METC142073
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2016-03

CONDITIONS: Anastomotic Leakage; Colorectal Cancer; Anastomotic Leak; Colorectal Neoplasms; Colorectal Carcinoma; Colorectal Tumors
Keywords: Colorectal carcinoma; Anastomotic leakage; Markers; Diagnosis
MeSH Terms: conditions — Anastomotic Leak; Colorectal Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swab for DNA Feces samples for microbiota analysis Blood serum for markers indicative of infection, ischemia/reperfusion injury or other Intestinal tissue from both ends of the resected colon segment Exhaled breath for VOCs collection and pattern analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Anastomotic leakage: Of the entire cohort, data collected from patients suffering from anastomotic leakage will be evaluated and compared to patients that did not develop anastomotic leakage. No interventions, only data collection.
  Interventions: Other: No interventions, only data collection
- No anastomotic leakage: Of the entire cohort, data collected from patients suffering from anastomotic leakage will be evaluated and compared to patients that did not develop anastomotic leakage. No interventions, only data collection.
  Interventions: Other: No interventions, only data collection

INTERVENTIONS:
Other: No interventions, only data collection — Only data is collected from the subjects in both groups.

SUMMARY:
Rationale: Colorectal cancer is the fourth most common cause of cancer death worldwide, estimated to be responsible for almost 610,000 deaths in 2008. Surgery remains the predominant curative treatment type for colorectal cancer, but has a major impact on the patient's wellbeing by demanding large amounts of metabolic reserves. This can lead to the development of frequently observed and severe postoperative complications. The most important complication after colorectal surgery is anastomotic leakage (AL), which has an incidence of 8-15% in the Netherlands. AL is associated with high short-term mortality rates of up to 40%. Even though many attempts have been made to reduce the incidence of this dreaded complication, none of these interventions have been successful so far. Despite proper patient selection and improvement in surgical techniques, the percentage of AL has been stable for years.

Objectives: To investigate whether recently identified patient-specific factors can predict the occurrence of anastomotic leakage in patients undergoing elective surgery for colorectal cancer.

Study design: Prospective observational study Study population: Adult colorectal cancer patients undergoing elective surgery. Main study parameters/endpoints: Primary endpoint: AL within 30 days postoperatively Secondary endpoints: Intestinal microbiome in fecal sample, I-FABP, SM22, Calprotectin, C-reactive protein(CRP), Citrullin, complement factors in blood, VOCs in exhaled air, COX-2 & MBL polymorphisms in buccal smear, L3-index & atherosclerosis measurements on CT-scans, SNAQ & MUST scores

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the fourth most common cause of cancer death worldwide, estimated to be responsible for 610,000 deaths in 20081. The number of CRC patients is concomitantly increasing due to a higher incidence, population growth, aging of the population and the recently established nationwide screening. Surgery remains the predominant curative treatment type for CRC, but has a major impact on the patient's wellbeing by demanding large amounts of metabolic reserves. This can lead to the development of frequently observed and severe postoperative complications. Anastomotic leakage (AL) is the most important complication after colorectal surgery and has an incidence of 8-15% in the Netherlands. AL is associated with high short-term mortality rates of up to 40%. Even though many attempts have been made to prevent this dreaded complication, none of these interventions have been successful so far. Despite proper patient selection, reduction of known preoperative risk factors and improved surgical techniques as well as introduction of 'fast track' protocol, AL incidence has not decreased in the past decade(s). AL is associated with a decreased disease-specific survival and an increased recurrence rate of CRC. The aim of this study is to investigate potential strategies to prevent AL, to be able to diagnose AL in time and therefore start treatment as early as possible in the process.

The etiology of anastomotic healing in the human gastrointestinal tract is not fully elucidated. Risk factors that are associated with anastomotic leakage have been identified, such as patient characteristics (age, malnutrition, tumor distally localized) and surgical factors (insufficient perfusion of the anastomosis, tension on the anastomosis).

Previous studies performed at our surgical research department of the School for Nutrition, Toxicology and Metabolism (NUTRIM) were focused on these risk factors individually. We revealed the consequences of intestinal ischemia both in small and large human intestines in a unique experimental model and described the recovery mechanism of the intestine after ischemic injury. The crucial role of Mannose Binding Lectin (MBL), an important complement factor of the immune system was shown as well as the fact that small proteins present in mature enterocytes (Intestinal-Fatty Acid Binding Proteins, I-FABP) can act as adequate markers in plasma for intestinal damage13-14. Furthermore, with the use of cyclooxygenase-2 (COX-2) knockout mice, it was shown that COX-2 is essential in the healing process of colonic anastomoses (manuscript submitted).

Another previous study showed that frailty (defined with the Groningen Frailty Index, sarcopenia (determined by measuring the skeletal muscle mass at L3 level at the CT-scan) and malnutrition (assessed with Short Nutritional Assessment Questionnaire (SNAQ) en Malnutrition Universal Screening Tool (MUST)) is associated with the occurrence of sepsis and mortality in 273 patients. In a pilot study with 90 patients, preoperative I-FABP plasma levels and postoperative inflammatory plasma concentration (C-reactive protein & calprotectin) were identified as predictive markers for anastomotic leakage after elective colorectal surgery. In addition, composition of volatile organic compounds (VOCs) in exhaled breath varies depending on health status. Various metabolic processes within the body produce volatile products that are released into the blood and will be passed on to the airway once the blood reaches the lungs. Moreover, the occurrence of chronic inflammation and/or oxidative stress can result in the excretion of volatile compounds that generate unique VOC patterns. In this study, we will measure the total amount of VOCs in exhaled air, to see if this is an eligible tool for early clinical diagnosis of anastomotic leakage.

Based on all these results, we aim to combine and translate observational results from individual studies into one multicentre prospective study in which several aspects of anastomotic leakage will be investigated. With the results of this study, we expect to be able to provide patients an adequate risk estimation regarding anastomotic leakage. This will help surgeons to make the decision to create a stoma instead of performing a primary anastomosis and to detect anastomotic leakage at an earlier stage. Furthermore, this study may provide new insights that can lead to potential new treatment.

ELIGIBILITY:
Inclusion Criteria:

* in need of laparoscopic or open large bowel resection with primary anastomosis as standard treatment for colorectal carcinoma

Exclusion Criteria:

* not requiring an anastomosis
* abdominal surgery in the past 4 weeks (with exception from temporary defunctioning ostomies for patients with obstructive colorectal tumours)
* pregnancy
* cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with colorectal cancer
Sampling Method: Probability Sample
Enrollment: 774 (Actual)
Dates: Start 2015-08; Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Anastomotic leakage | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Bouvy, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (4):
- Netherlands (4):
  - Zuyderland Medical Centre, Heerlen
  - Maastricht University Medical Centre, Maastricht
  - Zuyderland Medical Centre, Sittard
  - VieCuri Medical Centre, Venlo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jongen AC, Bosmans JW, Kartal S, Lubbers T, Sosef M, Slooter GD, Stoot JH, van Schooten FJ, Bouvy ND, Derikx JP. Predictive Factors for Anastomotic Leakage After Colorectal Surgery: Study Protocol for a Prospective Observational Study (REVEAL Study). JMIR Res Protoc. 2016 Jun 9;5(2):e90. doi: 10.2196/resprot.5477. PMID 27282451